CLINICAL TRIAL: NCT02743117
Title: A Phase 4 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of 1 New 6:2 Influenza Virus Reassortant in Adults
Brief Title: Study to Evaluate the Safety of 1 New 6:2 Influenza Virus Reassortant in Adults for the 2016-2017 Season
Acronym: FluMist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D2560C00012
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Influenza; Healthy
Keywords: Trivalent; Influenza; FluMist Quadrivalent; Vaccine; Prevention; Healthy; Monovalent
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monovalent Influenza Vaccine (Experimental): A single dose of 10^(7.0 +/- 0.5) fluorescent focus units (FFU) strain of monovalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Biological: Monovalent Influenza Vaccine
- Placebo (Placebo Comparator): A single dose of placebo matched to monovalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Monovalent Influenza Vaccine — A single dose of 10^(7.0 ± 0.5) FFU strain of monovalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Monovalent Influenza Vaccine
Other: Placebo — A single dose of placebo matched to monovalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study is designed to evaluate the safety of 1 new influenza virus vaccine strain to be included in FluMist Quadrivalent for the 2016-2017 influenza season

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age. Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of monovalent vaccine or placebo by intranasal spray. Randomization will be stratified by site. This study will be conducted at 3 sites in the United States of America. Each subject will receive 1 dose of investigational product on Day 1. The duration of study participation for each subject is the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 49 years
* Written informed consent
* Subject available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the Investigator

Exclusion Criteria:

* Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (example [eg], asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (greater than [>] 100.0 degrees Fahrenheit [F] oral or equivalent) and/or clinically significant respiratory illness (example, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, South Miami, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 301 participants were randomized and participated in the study from 02-May-2016 through 30-Nov-2016 at 3 sites in the United States of America (USA).
Pre-assignment Details: One participant was considered as screen failure and 300 randomized participants were treated in the study.
Groups:
- Placebo: Participants received a single dose of placebo matching with monovalent influenza vaccine by intranasal spray on Day 1.
- Monovalent Influenza Vaccine: Participants received a single dose of monovalent influenza vaccine [10^7.0 +/- 0.5 fluorescent focus unit (FFU) of each of 1 cold adapted (ca), attenuated (att), temperature sensitive (ts) 6:2 reassortant influenza strains] by intranasal spray on Day 1.
Period: Overall Study
Arm/Group | Placebo | Monovalent Influenza Vaccine
Started | 60 | 241
Treated | 59 | 241
Completed | 59 | 240
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants that were randomized and treated with investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Monovalent Influenza Vaccine | Total
Number analyzed (Participants) | 59 | 241 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.2 (9.4) | 33.3 (9.5) | 33.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 139 | 172
  Male | 26 | 102 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fever Greater Than or Equal to (>=) 101 Degrees Fahrenheit (F)
Description: Percentage of participants with fever defined as oral temperature >=101 degrees F were reported.
Time Frame: Baseline (Day 1) up to Day 8
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Monovalent Influenza Vaccine
Number analyzed (Participants) | 59 | 241
Percentage of participants | 1.7 | 0.4
Statistical Analysis 1: Comparison: Placebo vs Monovalent Influenza Vaccine; Test type: Superiority or Other; Rate Difference = -1.3, 95% CI 2-sided [-8.1 to 1.3]

2. Secondary Outcome: Percentage of Participants With Solicited Symptoms
Description: Solicited symptoms are predefined symptoms or events specifically inquired about and assessed daily after vaccine administration up to 15 days after vaccination. The solicited symptoms include fever greater than (>) 100.0 degrees F (37.8 degrees Celsius), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity and headache. Results were reported for all solicited symptoms except fever >=101 degrees F (reported as primary outcome) up to 8 days after vaccination and all solicited symptoms up to 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Monovalent Influenza Vaccine
Number analyzed (Participants) | 59 | 241
Percentage of participants
  Up to Day 8 | 33.9 | 25.7
  Up to Day 15 | 37.3 | 29.9
Statistical Analysis 1: Comparison: Placebo vs Monovalent Influenza Vaccine; Up to Day 8; Test type: Superiority or Other; Rate Difference = -8.2, 95% CI 2-sided [-22.2 to 4.6]
Statistical Analysis 2: Comparison: Placebo vs Monovalent Influenza Vaccine; Up to Day 15; Test type: Superiority or Other; Rate Difference = -7.4, 95% CI 2-sided [-21.6 to 5.9]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were events between administration of study drug and up to 15 days after vaccination that are absent before treatment or that worsened relative to pre-treatment state. Results were given for AEs reported up to 8 days and 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | Monovalent Influenza Vaccine
Number analyzed (Participants) | 59 | 241
Participants
  Up to Day 8 | 1 | 9
  Up to Day 15 | 1 | 14

4. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) and New Onset Chronic Diseases (NOCDs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs were serious events between administration of study drug and up to 181 days after the dose that are absent before treatment or that worsen relative to pretreatment state. An NOCD is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant. Results were given for TESAEs and NOCDs reported up to 29 days and 181 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 29 and Day 181
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | Monovalent Influenza Vaccine
Number analyzed (Participants) | 59 | 241
Participants
  Up to Day 29: TESAEs | 0 | 0
  Up to Day 29: NOCDs | 0 | 0
  Up to Day 181: TESAEs | 0 | 0
  Up to Day 181: NOCDs | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Require Antipyretic and/or Analgesic Medication
Description: Percentage of participants who require antipyretic and/or analgesic medication were reported.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Monovalent Influenza Vaccine
Number analyzed (Participants) | 59 | 241
Percentage of participants
  Up to Day 8 | 3.4 | 1.2
  Up to Day 15 | 5.1 | 1.7

ADVERSE EVENTS:
Time Frame: Adverse Events: From Screening (Day -14) up to Day 15, and Serious Adverse Events: From Screening (Day -14) up to Day 181
Arm/Group | Placebo | Monovalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/241
Other Adverse Events (participants affected / at risk) | 1/59 | 14/241
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | Monovalent Influenza Vaccine (N=241)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.